CLINICAL TRIAL: NCT00424515
Title: A Phase II Study of Imatinib in Patients With Mucosal or Acral/Lentiginous Melanoma and Melanomas That Arise on Chronically Sun Damaged Skin.
Brief Title: Imatinib in Patients With Mucosal or Acral/Lentiginous Melanoma
Acronym: BUS255
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, F. Stephen Hodi, MD, Melanoma Disease Center Director, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-056
Record Dates: First submitted 2007-01-18; First posted 2007-01-19 (Estimated); Results first posted 2016-12-08 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2016-06

CONDITIONS: Mucosal Melanoma; Acral/Lentiginous Melanoma; Chronically Sun Damaged Melanomas
Keywords: Imatinib; Gleevec
MeSH Terms: interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment Arm (Experimental): Imatinib
  Interventions: Drug: Imatinib

INTERVENTIONS:
Drug: Imatinib — Imatinib was given at a dose of 400 mg orally daily (4 100mg pills). Patients received treatment up to 12 months as long as they were receiving clinical benefit. Dosage may have been increased to twice daily if disease worsened and patient was in otherwise good clinical condition.
  Other Names: Gleevec

SUMMARY:
The purpose of this study is to evaluate how effective imatinib (Gleevec) is in treating acral/lentiginous and mucosal melanoma which has spread to other parts of the body in patients who's disease carries a c-kit mutation. Imatinib is a protein-kinase inhibitor. It is believed that imatinib may be effective in blocking signals on certain cancer cells which allow the malignant cells to multiply and spread.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the response rate of patients with metastatic mucosal, acral/lentiginous, or chronically sun damaged melanomas to treatment with of imatinib.
* To determine the time to progression.

Secondary

* To correlate c-kit mutational status with response to therapy.
* To evaluate the use of FDG-PET scanning in determining early biologic response to therapy.
* Tolerability of imatinib.
* To assess amplification of c-kit status through quantitative PCR and/or FISH and other related molecular pathway targets.
* To correlate c-kit amplification status with response to therapy.

ELIGIBILITY:
Inclusion Criteria:

* Melanomas that arise on chronically sun damaged skin and have pathologic evidence of solar elastosis
* History of primary mucosal or acral/lentiginous melanoma
* Histologically documented stage IV metastatic melanoma
* ECOG performance status 0,1, or 2
* Estimated life expectancy of 6 months or greater
* Age 18 years or older
* Creatinine < 1.5 x ULN
* ANC > 1500 ul
* Platelets > 100,000 ul
* Total bilirubin, AST, and ALT < 2 x ULN
* Amylase and lipase < 1.5 x ULN
* C-kit mutation documented from either primary or metastatic tumor site
* > 4 weeks from prior chemotherapy or investigational drug
* At least one measurable site of disease as defined by at least 1 cm in greatest dimension

Exclusion Criteria:

* Severe and/or uncontrolled medical disease
* Pregnant or nursing mothers
* Any other significant medical, surgical, or psychiatric condition that my interfere with compliance
* Patient is < 5 years free of another primary malignancy except: basal cell skin cancer or a cervical carcinoma in situ
* Concurrent treatment with Warfarin
* Prior treatment with c-kit inhibitor
* Patient with Grade III/IV cardiac problems as defined by NYHA criteria
* No H2 blockers or proton pump inhibitors
* Known brain metastasis
* Known chronic liver disease
* Known diagnosis of HIV infection
* Previous radiotherapy to > 25% of the bone marrow
* Major surgery within 2 weeks prior to study entry
* Patient has received any other investigational agent within 28 days of first study drug dosing
* Chemotherapy within 4 weeks prior to study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2006-07; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: F. Stephen Hodi, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (5):
- United States (5):
  - University of Colorado at Denver Health Sciences Center, Denver, Colorado
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - University of Chicago, Chicago, Illinois
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hodi FS, Corless CL, Giobbie-Hurder A, Fletcher JA, Zhu M, Marino-Enriquez A, Friedlander P, Gonzalez R, Weber JS, Gajewski TF, O'Day SJ, Kim KB, Lawrence D, Flaherty KT, Luke JJ, Collichio FA, Ernstoff MS, Heinrich MC, Beadling C, Zukotynski KA, Yap JT, Van den Abbeele AD, Demetri GD, Fisher DE. Imatinib for melanomas harboring mutationally activated or amplified KIT arising on mucosal, acral, and chronically sun-damaged skin. J Clin Oncol. 2013 Sep 10;31(26):3182-90. doi: 10.1200/JCO.2012.47.7836. Epub 2013 Jun 17. PMID 23775962
- [Derived] Zukotynski K, Yap JT, Giobbie-Hurder A, Weber J, Gonzalez R, Gajewski TF, O'Day S, Kim K, Hodi FS, Van den Abbeele AD. Metabolic response by FDG-PET to imatinib correlates with exon 11 KIT mutation and predicts outcome in patients with mucosal melanoma. Cancer Imaging. 2014 Nov 12;14(1):30. doi: 10.1186/s40644-014-0030-0. PMID 25609545

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was activated on July 6, 2006 and closed March 1, 2011. Patients enrolled from 9 medical centers beginning April 2007 through December 2010.
Groups:
- Amplified KIT; Mutated KIT: Imatinib was given at a dose of 400 mg orally daily (4 100 mg pills). Patients received treatment up to 12 months as long as they were receiving clinical benefit. Dosage may have been increased to twice daily if disease worsened and patient was in otherwise good clinical condition. Patients were classified into two cohorts based upon KIT molecular status.
Period: Overall Study
Arm/Group | Amplified KIT | Mutated KIT
Started | 11 | 13
Completed | 0 | 0
Not Completed | 11 | 13
Not completed — Progressive Disease | 10 | 11
Not completed — Adverse Event | 0 | 1
Not completed — Intercurrent Illness | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: The analysis dataset is comprised of enrolled and treated patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | Amplified KIT | Mutated KIT | Total
Number analyzed (Participants) | 11 | 13 | 24
Age, Continuous [Median (Full Range); unit: years] | 69 [55 to 84] | 64 [42 to 80] | 65 [42 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 11 | 18
  Male | 4 | 2 | 6
Region of Enrollment [Number; unit: participants]
  United States | 11 | 13 | 24
Melanoma Type [Number; unit: participants]
  Acral | 4 | 2 | 6
  Mucosal | 6 | 11 | 17
  Chronically Sun-Damaged | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Best Overall Response
Description: Best overall response (BOR) on treatment was based on RECIST 1.0 criteria. For target lesions, complete response (CR) is complete disappearance of all target lesions and partial response (PR) is at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD. CR or PR confirmation required within 4 weeks. Progressive disease (PD) is at least a 20% increase in the sum LD of target lesions from smallest sum LD as reference or the appearance of one or more new lesions. Stable disease (SD) is neither meeting PR or PD. PD for the evaluation of non-target lesions is the appearance of one or more new lesions and/or unequivocal progression of non-target lesions. CR is disappearance of all non-target lesions.
Time Frame: Disease was evaluated radiologically at baseline, after 6-weeks, and at 2-month intervals on treatment. Mean treatment duration was 4 months (range 1-11; amplified/mutated 3m/ 6m).
Population: The analysis dataset is comprised of treated patients.
Measure: Number; unit: participants
Arm/Group | Amplified KIT | Mutated KIT
Number analyzed (Participants) | 11 | 13
participants
  Complete Response | 0 | 0
  Partial Response | 0 | 7
  Stable Disease | 2 | 3
  Progressive Disease | 9 | 3

2. Secondary Outcome: Time to Progression
Description: Time to progression (TTP) based on the Kaplan-Meier method is defined as the duration of time from study entry to documented disease progression (PD) requiring removal from the study. Per RECIST 1.0 criteria: progressive disease (PD) is at least a 20% increase in the sum of longest diameter (LD) of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. PD for the evaluation of non-target lesions is the appearance of one or more new lesions and/or unequivocal progression of non-target lesions.
Time Frame: Disease was evaluated radiologically at baseline, after 6-weeks, and at 2-month intervals on treatment and every 3 months long-term. Mean treatment duration was 4 months (range 1-11; amplified/mutated 3m/ 6m).
Population: The analysis dataset is comprised of treated patients.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Amplified KIT | Mutated KIT
Number analyzed (Participants) | 11 | 13
months | 3.4 [1.0 to 5.7] | 3.9 [2.6 to 6.6]

3. Secondary Outcome: Overall Survival
Description: Overall survival (OS) is defined as the time from study entry to death or date last known alive.
Time Frame: Patients were followed long-term every 3 months until first progression, death or lost to follow-up. Median survival follow-up was 10.6 months (range 3.7-27.1).
Population: The analysis dataset is comprised of treated patients.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Amplified KIT | Mutated KIT
Number analyzed (Participants) | 11 | 13
months | 11.9 [4.5 to 16.2] | 12.9 [5.5 to 24.3]

ADVERSE EVENTS:
Time Frame: AE assessment occurred every other month from the start of study drug and up to day 30 post-treatment.
Description: Maximum grade toxicity by type was first calculated. Serious AEs were defined as events with treatment-attribution of possibly, probably or definitely and grade 3 or higher per CTCAEv3. Other AEs were defined as events with treatment-attribution of possible, probable or definite and grades 1 or 2 per CTCAEv3.
Arm/Group | Amplified KIT | Mutated KIT
Serious Adverse Events (participants affected / at risk) | 1/11 | 3/13
Other Adverse Events (participants affected / at risk) | 9/11 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Amplified KIT (N=11) | Mutated KIT (N=13)
Hemoglobin (Blood and lymphatic system disorders) | 0 | 2
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1
Leukocytes (Investigations) | 0 | 1
Lymphopenia (Investigations) | 1 | 1
Neutrophils (Investigations) | 0 | 1
Pruritus/itching (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Amplified KIT (N=11) | Mutated KIT (N=13)
Abdomen, pain (Gastrointestinal disorders) | 0 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1
ALT, SGPT (Investigations) | 0 | 2
Anorexia (Metabolism and nutrition disorders) | 3 | 2
AST, SGOT (Investigations) | 0 | 3
Bicarbonate (Metabolism and nutrition disorders) | 0 | 1
Bilirubin (Investigations) | 1 | 0
Bruising (Injury, poisoning and procedural complications) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 2
Constitutional (General disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Creatinine (Investigations) | 1 | 1
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 2 | 7
Distention/bloating, abdominal (Gastrointestinal disorders) | 0 | 1
Dizziness (Nervous system disorders) | 2 | 2
Dry mouth (Gastrointestinal disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Edema head and neck (General disorders) | 1 | 6
Edema limb (General disorders) | 0 | 7
Edema trunk/genital (General disorders) | 0 | 1
Fatigue (General disorders) | 7 | 7
Flatulence (Gastrointestinal disorders) | 0 | 2
Flu-like syndrome (General disorders) | 0 | 1
Flushing (Vascular disorders) | 0 | 1
GI (Gastrointestinal disorders) | 1 | 3
Glomerular filtration rate (Renal and urinary disorders) | 0 | 1
Head/headache (Nervous system disorders) | 1 | 0
Hematologic (Blood and lymphatic system disorders) | 0 | 1
Hemoglobin (Blood and lymphatic system disorders) | 3 | 3
Hemoglobinuria (Renal and urinary disorders) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1
Hypernatremia (Metabolism and nutrition disorders) | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 2
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1
Leukocytes (Investigations) | 2 | 1
Lymphatics (Blood and lymphatic system disorders) | 1 | 0
Metabolic/Laboratory (Investigations) | 1 | 1
Nausea (Gastrointestinal disorders) | 4 | 8
Neutrophils (Investigations) | 2 | 2
Ocular (Eye disorders) | 0 | 1
Optic disc edema (Eye disorders) | 0 | 1
Platelets (Investigations) | 0 | 1
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pruritus/itching (Skin and subcutaneous tissue disorders) | 1 | 3
Pulmonary/Upper Respiratory (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rash/desquamation (Skin and subcutaneous tissue disorders) | 0 | 4
Rigors/chills (General disorders) | 1 | 1
Skin (Skin and subcutaneous tissue disorders) | 0 | 1
Sweating (Skin and subcutaneous tissue disorders) | 0 | 2
Taste disturbance (Nervous system disorders) | 3 | 1
Tearing (Eye disorders) | 1 | 1
Tremor (Nervous system disorders) | 0 | 1
Ulceration (Skin and subcutaneous tissue disorders) | 0 | 1
Vascular (Vascular disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 4
Weight loss (Investigations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No